CLINICAL TRIAL: NCT03651830
Title: A Prosthetic Foot Emulator to Optimize Prescription of Prosthetic Feet in Veterans and Service Members With Leg Amputations
Brief Title: A Test-Drive Strategy for the Prescription of Prosthetic Feet for People With Leg Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); Stanford University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MD13; W81XWH-16-1-056 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-08-15; First posted 2018-08-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Amputation
Keywords: Amputation; Rehabilitation; Prescriptions; Emulator; Prosthetics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prosthetic Foot Emulator (Experimental): The Prosthetic Foot Emulator (PFE) is a customizable robotic prosthetic foot that can mimic commercial feet to predict how individual patients will respond to candidate feet. Participants will walk with the PFE using three different modes (emulating three commercial feet) under different walking conditions.
  Interventions: Device: Prosthetic Foot Emulator
- Commercially available prosthetic feet (Active Comparator): Participants will walk under different walking conditions using three different commercial prosthetic feet.
  Interventions: Device: Commercially available prosthetic feet

INTERVENTIONS:
Device: Prosthetic Foot Emulator — Participants will walk in the laboratory with the Prosthetic Foot Emulator (PFE) in three foot modes corresponding to actual study feet. Walking conditions will include self-selected speed, slow speed, fast speed, incline, and up stairs.
  Arms: Prosthetic Foot Emulator
Device: Commercially available prosthetic feet — Participants will walk in the laboratory with three different commercially available prosthetic feet. Walking conditions will include self-selected speed, slow speed, fast speed, incline, and up stairs.
  Additionally, participants will be fit with one of the actual feet and wear it at home and in the community for approximately two weeks. This will be followed by two-week periods in the community with each of the other two commercially available prosthetic feet.
  Arms: Commercially available prosthetic feet

SUMMARY:
Objective/Hypotheses and Specific Aims: The primary aim of this proposal is to determine whether a PFE can be used to predict foot preference and mobility outcomes with corresponding commercial prosthetic feet in people with a unilateral transtibial amputation (TTA). Secondarily, the investigators aim to determine whether a brief trial of commercial prosthetic feet would be able to similarly predict longer-term foot preference and mobility outcomes with those feet.

Study Design: The investigators will use a participant blinded cross-over study with repeated measurements. Participants with TTA will be enrolled at each of the three study sites: two VA sites (Puget Sound and Minneapolis), and one Department of Defense site (Center for the Intrepid). Participants will complete up to 6 visits. After an initial assessment visit, participants will be assigned to the high or low mobility group, and then during visit 2 they will be randomized to use the PFE in three foot modes or the three corresponding actual (commercially available) feet during walking tests in the laboratory. During visit 3 participants will repeat the procedures in the other condition (e.g., PFE if Day 2 included actual feet testing). At the end of visit 3 participants will be fit with one of the actual feet and wear it at home and in the community for approximately two weeks. At visit 4 participants will be fit with the next actual foot and repeat the 2 week use window. The same process will be followed for the final foot at visit 5, and the study foot will be returned at visit 6. Participants' preference, satisfaction and perceived mobility, and functional mobility will be measured and compared across all foot conditions (emulated and actual). After participants complete the procedures detailed above, they may be eligible to be invited to participate in follow-up phone interviews. A subset of participants may also be invited to participate in follow-up biomechanical data collection comparing the PFE foot conditions to the respective actual prosthetic feet during walking. Additionally, a subset of participants may also be invited to participate in follow-up data collection comparing prosthetic foot conditions of different stiffness categories.

DETAILED DESCRIPTION:
Objectives and Rationale: Using a prosthesis allows many who experience lower leg amputation to regain functional abilities, but walking may be more difficult, and a sub-optimal prosthesis can substantially restrict participation in desired activities. Selecting an optimal prosthetic foot is an important aspect of maximizing mobility and the achievement of functional goals for people with lower leg amputation, however there is limited evidence to guide this process. The current prosthetic prescription process relies on clinician experience and typically does not allow people with a leg amputation to easily try out different prosthetic feet. The investigators have developed a customizable robotic prosthetic foot that mimics the mechanical properties of commercially available prosthetic feet without physically changing feet. This 'prosthetic foot emulator' (PFE) can be attached to the prescribed prosthetic socket and worn like a regular prosthetic foot within the laboratory or clinic, providing people with leg amputations the opportunity to quickly 'test-drive' many prosthetic foot designs within a single test session. Trial and error with actual commercial prosthetic feet can be inefficient given the time and expense required for the purchasing and fitting of prosthetic feet. The PFE could provide a means to explore a range of feet in a very short period of time. This study will evaluate the ability of the emulator to accurately reproduce the experience of wearing several commercially available (actual) prosthetic feet. The investigators will test whether brief in-laboratory experiences with emulated or actual feet can accurately predict longer-term foot preference, satisfaction, and walking ability in the community. The investigators will also evaluate the experiences of prosthetic foot prescription practices using qualitative methods from follow-up phone interviews with participants. Finally, the investigators will evaluate biomechanical outcomes during walking between the PFE and actual prosthetic feet to examine the ability of the emulator to accurately reproduce the experience of walking with the actual feet. Results from this study may provide evidence to support a new approach to prosthesis prescription and could resolve longstanding uncertainty in the prescription process for prosthetic feet.

ELIGIBILITY:
Inclusion Criteria:

* has a unilateral (one leg) transtibial (below-knee) amputation
* has used a prosthetic limb for walking for at least six months
* has a comfortably fitting prosthetic socket
* be able to walk with a prosthetic limb sufficiently to participate in the experiment walking trials
* be age 18 to 89 years

Exclusion Criteria:

* contralateral limb or upper limb amputation
* are unable to use test feet for any reason (e.g., excessively long residual limb that is not compatible with wearing study prosthetic feet)
* unable to walk under the minimal necessary study walking conditions in order to complete the study procedures without undo stress
* currently pregnant (determined via self-report during screening)
* current surgical, neurological, rheumatologic, or lower limb musculoskeletal problem that significantly impairs ambulation (e.g., current ulcer, terminal illness, lower extremity joint replacement)
* weight greater than 250lbs.
* inadequate cognitive or language function to consent to participate
* currently incarcerated

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Foot Preference Survey | Administered during initial testing with prosthetic foot emulator (approximately 2 hours).
  Self-report survey related to prosthetic foot preference, satisfaction, and perceived mobility, with questions answered on 0-10 scale.
Foot Preference Survey | Administered during initial testing with actual prosthetic feet (approximately 2 hours).
  Self-report survey related to prosthetic foot preference, satisfaction, and perceived mobility, with questions answered on 0-10 scale.
Foot Preference Survey | Administered at 2-week follow up for prosthetic foot A.
  Self-report survey related to prosthetic foot preference, satisfaction, and perceived mobility, with questions answered on 0-10 scale.
Foot Preference Survey | Administered at 2-week follow up for prosthetic foot B.
  Self-report survey related to prosthetic foot preference, satisfaction, and perceived mobility, with questions answered on 0-10 scale.
Foot Preference Survey | Administered at 2-week follow up for prosthetic foot C.
  Self-report survey related to prosthetic foot preference, satisfaction, and perceived mobility, with questions answered on 0-10 scale.

SECONDARY OUTCOMES:
Two Minute Walk Test | Administered at baseline and at 2-week follow up for each foot condition.
  Participants are asked to walk for 2 minutes at their fastest possible speed and distance walked is recorded.
Prosthetic Limb Users Survey of Mobility (PLUS-M), tailored short-form | Administered at baseline and at 2-week follow up for each foot condition.
  Standardized self-report item bank.
Activities Specific Balance Confidence Scale (ABC) | Administered at baseline and at 2-week follow up for each foot condition.
  This is a subjective measure of confidence in performing ambulatory activities without falling or feeling unsteady. The investigators are using a revised version of the ABC recommended to ease administration and improve scoring. Questions answered on 0-4 scale (0 = No Confidence; 4 = Complete Confidence). Scores for 16 questions combined and averaged.
Trinity Amputation and Prosthesis Experience Scales (TAPES) | Administered at baseline and at 2-week follow up for each foot condition.
  Multidimensional health instrument that measures self-reported activity restrictions (TAPES-AR) and satisfaction with the function (TAPES-FUN) of a prosthesis. Other subscales of TAPES will not be used. Questions answered on 0-2 scale (0 = No, not limited; 2 = Yes, limited a lot for TAPES-AR, and 0= Not satisfied; 2 = Very satisfied for TAPES-FUN). Subscales will be scored separately. For TAPES-AR, scores of all items answered will be combined and averaged. For TAPES-FUN, scores for all items will be added together.
Four Square Step Test (FSST) | Administered at baseline and at 2-week follow up for each foot condition.
  Participants are asked to step over canes in a specific sequence as quickly as possible and two trials are timed and recorded.
Timed Up and Go (TUG) | Administered at baseline and at 2-week follow up for each foot condition.
  Participants are asked to start at sitting, stand and walk around a cone, and return to a seated position. Two trials are performed at both a comfortable pace and at a fast pace. All trials are timed and times are recorded.
Narrowing Beam Walking Test (NBWT) | Administered at baseline and at 2-week follow up for each foot condition.
  Participants are asked to walk as far as possible along a narrowing beam without using arms or assistance for balance. Five trails are completed and distances are recorded.
Berg Balance Scale (BBS) | Administered at baseline and at 2-week follow up for each foot condition.
  Participants are asked to perform a variety of tasks such as sitting, standing, turning, and transferring between chairs, in order to measure balance.
Kinematic and kinetic outcome analysis | up to 100 weeks
  Some participants are asked to complete biomechanical gait analysis while walking with the PFE and the corresponding actual prosthetic feet while wearing reflective markers in a motion capture laboratory (Vicon motion capture system). Ankle, knee, hip, trunk, and upper body motion data will be collected while participants walk at self-selected speeds on an instrumented treadmill. These kinematic and kinetic outcome data will be collected at follow-up study visits up to 100 weeks after enrollment and after participants complete previous study activities (note: only a subset of participants).

CONTACTS AND LOCATIONS:
Overall Officials: David Morgenroth, MD, Principal Investigator — VA Puget Sound Health Care System and SIBCR
Locations (3):
- United States (3):
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Center for the Intrepid, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No